CLINICAL TRIAL: NCT01181895
Title: A Randomized, Double-blind, Double-dummy, Parallel-group, Placebo Controlled (on Inhaled Corticosteroid Medication), Multicenter Study to Evaluate the Efficacy and Safety of Vilanterol Inhalation Powder (GW642444) and Salmeterol, Compared With Placebo in the Treatment of Persistent Asthma in Adults and Adolescents Uncontrolled on Inhaled Corticosteroids
Brief Title: Study B2C112060: A Study of the Efficacy and Safety of Vilanterol Inhalation Powder in Adults and Adolescents With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112060
Record Dates: First submitted 2010-07-15; First posted 2010-08-13 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vilanterol (Experimental): Vilanterol inhalation powder once daily + Placebo inhalation powder via Diskus twice daily for 12 weeks
  Interventions: Drug: Vilanterol; Drug: Placebo Inhalation Powder Diskus
- Salmeterol (Active Comparator): Placebo inhalation powder via NDPI once daily + Salmeterol inhalation powder twice daily for 12 weeks
  Interventions: Drug: Salmeterol Inhalation Powder; Drug: Placebo Inhalation Powder NDPI
- Placebo (Placebo Comparator): Placebo inhalation powder via NDPI once daily + Placebo inhalation powder via Diskus twice daily for 12 weeks
  Interventions: Drug: Placebo Inhalation Powder NDPI; Drug: Placebo Inhalation Powder Diskus

INTERVENTIONS:
Drug: Vilanterol — Vilanterol inhalation powder inhaled orally once daily for 12 weeks
  Arms: Vilanterol
Drug: Salmeterol Inhalation Powder — Salmeterol inhalation powder inhaled orally twice daily for 12 weeks
  Arms: Salmeterol
Drug: Placebo Inhalation Powder NDPI — Placebo inhalation powder inhaled orally via Novel Dry Powder Inhaler
  Arms: Placebo; Salmeterol
Drug: Placebo Inhalation Powder Diskus — Placebo inhalation powder inhaled orally twice daily for 12 weeks
  Arms: Placebo; Vilanterol

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of vilanterol inhalation powder administered once daily in the evening in adolescent and adult subjects 12 years of age and older with persistent asthma over a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient at least 12 years of age
* Both genders; females of childbearing potential must be willing to use birth control method
* Clinical diagnosis of asthma for ≥12 weeks
* Best pre-bronchodilator FEV1 of 40%-90% predicted
* Reversibility of FEV1 of at least 12% and 200mls
* Current asthma therapy that include an inhaled corticosteroid for at least 12 weeks prior to 1st visit
* Ability to use replace current short-acting rescue treatment with albuterol and ability to withhold albuterol use for at least 6 hours prior to study visits

Exclusion Criteria:

* History of life-threatening asthma
* Respiratory infection within last 4 weeks leading to change in asthma management
* Asthma exacerbation within last 3 months
* Concurrent respiratory disease or other disease that would confound study participation or affect subject safety
* Allergies to study drugs, study drugs' excipients, or medications related to study drugs
* Taking another investigational medication or medication prohibited for use during the study.
* Previous participation in a vilanterol (GW642444) study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2010-09-01; Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (11):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Chester, South Carolina
  - GSK Investigational Site, Clinton, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
- Germany (4):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- Peru (5):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Isidro, Lima region
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Callao, Lima
  - GSK Investigational Site, Lima
- Poland (3):
  - GSK Investigational Site, Chrzanów
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Yalta

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lotvall J, Bateman ED, Busse WW, O'Byrne PM, Woodcock A, Toler WT, Jacques L, Goldfrad C, Bleecker ER. Comparison of vilanterol, a novel long-acting beta2 agonist, with placebo and a salmeterol reference arm in asthma uncontrolled by inhaled corticosteroids. J Negat Results Biomed. 2014 Jun 13;13(1):9. doi: 10.1186/1477-5751-13-9. PMID 24928338
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112060 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 347 participants (par.) were randomized to treatment; all 347 were included in the Intent-to-Treat (ITT) Population. One par. was not randomized but received treatment in error. This par. was not included in the ITT Population and is thus not captured in the Participant Flow module. This par. is categorized as being enrolled in the study (n=348).
Pre-assignment Details: Participants (par.) meeting eligibility criteria at the Screening visit completed a 28-day Run-in Period for Baseline, safety evaluations, and measures of asthma status. Par. were then randomized to an 8-week Treatment Period. A total of 583 par. were screened, and 347 were randomized, of which 298 received at least one dose of study treatment.
Groups:
- Placebo: Participants received placebo once daily (OD) in the evening from the dry powder inhaler (DPI) and placebo twice daily (BID) from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 12 weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study.
- Vilanteral 25 µg OD: Participants received Vilanterol (VI) 25 micrograms (µg) OD in the evening from the DPI and placebo BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) for 12 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
- Salmeterol 50 µg BID: Participants received Salmeterol 50 µg BID from the DISKUS/ACCUHALER (one inhalation in the morning and one inhalation in the evening) plus placebo OD in the evening from the DPI for 12 weeks. In addition, participants were provided supplemental albuterol/salbutamol aerosol to be used as needed throughout the study.
Period: Overall Study
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Started | 116 | 115 | 116
Completed | 99 | 101 | 98
Not Completed | 17 | 14 | 18
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Lack of Efficacy | 8 | 9 | 9
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Investigator Discretion | 1 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID | Total
Number analyzed (Participants) | 116 | 115 | 116 | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (16.64) | 41.0 (17.81) | 41.1 (16.84) | 41.3 (17.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 68 | 77 | 204
  Male | 57 | 47 | 39 | 143
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 11 | 5 | 6 | 22
  American Indian or Alaska Native | 37 | 44 | 41 | 122
  Japanese/East Asian Heritage | 0 | 0 | 1 | 1
  White | 68 | 66 | 68 | 202

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted-mean 24-hour Serial Forced Expiratory Volume in One Second (FEV1) at Week 12
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forcefully exhaled in one second. The weighted mean is calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5, 15, and 30 minutes (min) and at 1, 2, 3, 4, 11, 12, 12.5, 13, 14, 16, 20, 23, and 24 hours, respectively, at Week 12. The Baseline value was the Day 1 pre-dose FEV1 measurement. Change from Baseline is calculated as the weighted mean 0-24 hour FEV1 (Liters) at Week 12 minus the Baseline value. Analysis was performed using analysis of covariance (ANCOVA) with covariates of Baseline FEV1, region, sex, age, and treatment.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 95 | 101 | 100
Liters | 0.289 (0.0429) | 0.359 (0.0416) | 0.283 (0.0419)
Statistical Analysis 1: Comparison: Placebo vs Vilanteral 25 µg OD; Test type: Superiority or Other; p = 0.244, ANCOVA — P-value for the adjusted treatment difference for Vilanterol 25 µg OD versus Placebo; Mean Difference (Final Values) = 0.070, 95% CI 2-sided [-0.048 to 0.188] — The estimated value represents the adjusted treatment difference in the weighted mean 0-24 hour FEV1 (Liters) at Week 12 for Vilanterol 25 µg OD versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Salmeterol 50 µg BID; Test type: Superiority or Other; p = 0.926, ANCOVA — P-value for the adjusted treatment difference for Salmetarol 50 µg BID versus Placebo; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.124 to 0.113] — The estimated value represents the adjusted treatment difference in the weighted mean 0-24 hour FEV1 (Liters) at Week 12 for Salmeterol 50 µg BID versus Placebo

2. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: The time span during which the participants did not have to take any rescue bronchodilator (medication intended to relieve symptoms immediately) was considered to be a rescue-free period. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant (including the day of randomization). Change from Baseline is calculated as the value at Weeks 1-12 minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 115 | 115 | 114
Percentage of rescue-free 24-hr periods | 14.6 (2.71) | 21.7 (2.68) | 22.9 (2.72)

3. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: Participants who were symptom free for 24-hour periods during the12-week treatment period were assessed. The Baseline value was derived from the last 7 days of the daily diary prior to the randomization of the participant (including the day of randomization). Change from Baseline is calculated as the value at Weeks 1-12 minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 115 | 115 | 114
Percentage of symptom-free 24-hr periods | 12.7 (2.58) | 19.4 (2.55) | 19.5 (2.59)

4. Secondary Outcome: Change From Baseline in Individual Serial FEV1 Assessments at the End of the 12-week Treatment Period, Including the 12-hour and 24-hour Time Points
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forcefully exhaled in one second. The individual serial FEV1 is calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5, 15, 30, and 60 minutes (min) and 2, 3, 5, 11, 12, 12.5, 13, 14, 16, 20, 23, and 24 hours, relatively, on Treatment Day 84 (Week 12). The Baseline value was the Day 1 pre-dose FEV1 measurement. Change from Baseline was calculated as the value of the individual serial FEV1 taken at Week 12 minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline FEV1, region, sex, age, and treatment. Analysis was performed separately for each planned time point.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 116 | 115 | 116
Liters
  Predose, n=97,104,101 | 0.302 (0.0446) | 0.272 (0.0430) | 0.233 (0.0437)
  5 min, n=95,100,98 | 0.313 (0.0450) | 0.301 (0.0438) | 0.214 (0.0443)
  15 min, n=96, 101, 99 | 0.308 (0.0450) | 0.324 (0.0439) | 0.257 (0.0444)
  30 min, n=,96,101,100 | 0.322 (0.0443) | 0.344 (0.0432) | 0.272 (0.0435)
  60 min, n=96, 101, 100 | 0.336 (0.0445) | 0.352 (0.0433) | 0.296 (0.0437)
  2 hours, n=96, 100, 99 | 0.313 (0.0455) | 0.369 (0.0446) | 0.335 (0.0449)
  3 hours, n=96, 101, 100 | 0.304 (0.0455) | 0.374 (0.0444) | 0.316 (0.0447)
  4 hours, n=96, 101, 100 | 0.311 (0.0450) | 0.359 (0.0438) | 0.293 (0.0441)
  5 hours, n=96, 100, 100 | 0.292 (0.0455) | 0.368 (0.0445) | 0.279 (0.0447)
  11 hours, n=94, 99, 96 | 0.195 (0.0508) | 0.312 (0.0494) | 0.179 (0.0505)
  12 hours, n=93,98,95 | 0.250 (0.0477) | 0.341 (0.0465) | 0.217 (0.0473)
  12.5 hours, n=96, 97, 98 | 0.270 (0.0446) | 0.337 (0.0444) | 0.282 (0.0443)
  13 hours, 96, 98, 100 | 0.312 (0.0448) | 0.341 (0.0442) | 0.304 (0.0440)
  14 hours, n=95, 99, 99 | 0.341 (0.0445) | 0.401 (0.0436) | 0.359 (0.0437)
  16 hours, n=95, 98, 97 | 0.364 (0.0464) | 0.371 (0.0457) | 0.357 (0.0461)
  20 hours, n= 94, 101, 99 | 0.318 (0.0485) | 0.371 (0.0467) | 0.296 (0.0473)
  23 hours, 94, 101, 99 | 0.310 (0.0456) | 0.345 (0.0440) | 0.271 (0.0446)
  24 hours, n= 95, 101, 100 | 0.301 (0.0445) | 0.330 (0.0432) | 0.275 (0.0435)

5. Secondary Outcome: Change From Baseline in Daily Trough (Pre-dose and Pre-rescue Bronchodilator) PM (Evening) Peak Expiratory Flow (PEF) Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Trough PEF is the PEF measured approximately 24 hours after the last administration of study drug. The Baseline value is the average value of the last 7 days of daily PM PEF prior to randomization. Change from Baseline in trough PM PEF was calculated as the averaged value of all daily PM PEF for Week 1 to Week 12 minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute (L/min)
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 115 | 115 | 114
Liters per minute (L/min) | 11.0 (3.15) | 24.9 (3.14) | 18.8 (3.17)

6. Secondary Outcome: Change From Baseline in Daily AM (Morning) PEF Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Trough PEF is the PEF measured approximately 24 hours after the last administration of study drug. The Baseline value is the average value of the last 7 days of daily AM PEF prior to randomization. Change from Baseline in trough AM PEF was calculated as the averaged value of all daily AM PEF for Weeks 1 to Week 12 minus the value at Baseline. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute (L/min)
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 115 | 115 | 114
Liters per minute (L/min) | 14.2 (3.25) | 28.0 (3.24) | 23.6 (3.27)

7. Secondary Outcome: Number of Participants With the Indicated Time to an Increase of >=12% and >=200 Milliliters (mL) Above Baseline in FEV1 on Day 1 and Day 84 (0-2 Hours)
Description: The number of participants with a >=12% and >=200 mL increase from Baseline in FEV1 (the maximal amount of air that can be forcefully exhaled in one second) was evaluated on Day 1 and Week 12 for the time to a >=12% increase from Baseline (at the 5 minutes (min), 15 min, 30 min, 1hour (hr), and 2 hr nominal time points. Participants who did not achieve a >=12% and >=200 mL increase from Baseline in FEV1 over this time period were considered censored.
Time Frame: Day 1 and Week 12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 113 | 115 | 116
Participants
  Day 1, 5 min, n=113, 115, 116 | 23 | 33 | 18
  Day 1, 15 min, n=113, 115, 116 | 2 | 11 | 11
  Day 1, 30 min, n=113, 115, 1116 | 3 | 8 | 13
  Day 1, 1 hr, n=113, 115, 116 | 3 | 7 | 6
  Day 1, 2 hr, n=113, 115, 116 | 5 | 6 | 11
  Day 1, Censored, n=113, 115, 116 | 77 | 50 | 57
  Week 12, 5 min, n=96, 101, 100 | 39 | 42 | 30
  Week 12, 15 min, n=96, 101, 100 | 6 | 2 | 7
  Week 12, 30 min, n=96, 101, 100 | 2 | 2 | 8
  Week 12, 1 hr, n=96, 101, 100 | 1 | 4 | 5
  Week 12, 2 hr, n=96, 101, 100 | 3 | 7 | 4
  Week 12, Censored, n=96, 101, 100 | 45 | 44 | 46

8. Secondary Outcome: Number of Participants With the Indicated Global Assessment of Change Questionnaire Responses at the End of Week 4 and Week 12
Description: At the end of Week 4 and Week 12, the Global Assessment of Change Questionnaire, which assesses changes in asthma symptoms and rescue medication use, was completed by participants using the following scale: asthma symptom (AS) change: much better, somewhat better, a little better, the same, a little worse, somewhat worse, much worse; rescue medication use (RMU): much less often , somewhat less often , a little less often , the same , a little more often , somewhat more often , much more often.
Time Frame: Week 4 and Week 12
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Number analyzed (Participants) | 110 | 109 | 110
Participants
  Week 4, AS: Much better, n=110, 109, 110 | 25 | 37 | 34
  Week 4, AS: Somewhat better, n=110, 109, 110 | 35 | 43 | 34
  Week 4, AS: A little better, n=110, 109, 110 | 24 | 14 | 21
  Week 4, AS: The same, n=110, 109, 110 | 17 | 13 | 16
  Week 4, AS: A little worse, n=110, 109, 110 | 6 | 1 | 3
  Week 4, AS: Somewhat worse, n=110, 109, 110 | 2 | 0 | 2
  Week 4, AS: Much worse, n=110, 109, 110 | 1 | 1 | 0
  Week 4, RMU: Much less often, n=110, 109, 110 | 18 | 33 | 28
  Week 4, RMU: Somewhat less often, n=110, 109, 110 | 40 | 31 | 36
  Week 4, RMU: A little less often, n=110, 109, 110 | 18 | 23 | 20
  Week 4, RMU: The same, n=110, 109, 110 | 26 | 18 | 17
  Week 4, RMU: A little more often, n=110, 109, 110 | 4 | 3 | 7
  Week 4, RMU: Somewhat more often, n=110, 109, 110 | 2 | 0 | 2
  Week 4, RMU: Much more often, n=110, 109, 110 | 2 | 1 | 0
  Week 12, AS: Much better, n=100, 105, 101 | 31 | 52 | 35
  Week 12, AS: Somewhat better, n=100, 105, 101 | 35 | 31 | 34
  Week 12, AS: A little better, n=100, 105, 101 | 13 | 9 | 16
  Week 12, AS: The same, n=100, 105, 101 | 12 | 9 | 11
  Week 12, AS: A little worse, n=100, 105, 101 | 4 | 2 | 4
  Week 12, AS: Somewhat worse, n=100, 105, 101 | 4 | 1 | 1
  Week 12, AS: Much worse, n=100, 105, 101 | 1 | 1 | 0
  Week 12, RMU: Much less often, n=100, 105, 101 | 25 | 40 | 32
  Week 12, RMU: Somewhat less often, n=100, 105, 101 | 31 | 32 | 29
  Week 12, RMU: A little less often, n=100, 105, 101 | 13 | 16 | 13
  Week 12, RMU: The same, n=100, 105, 101 | 23 | 11 | 21
  Week 12, RMU: A little more often, n=100, 105, 101 | 2 | 5 | 4
  Week 12, RMU: Somewhat more often, n=100, 105, 101 | 4 | 0 | 2
  Week 12, RMU: Much more often, n=100, 105, 101 | 2 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Vilanteral 25 µg OD | Salmeterol 50 µg BID
Serious Adverse Events (participants affected / at risk) | 1/116 | 1/115 | 0/116
Other Adverse Events (participants affected / at risk) | 26/116 | 26/115 | 21/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=116) | Vilanteral 25 µg OD (N=115) | Salmeterol 50 µg BID (N=116)
Sudden death (General disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=116) | Vilanteral 25 µg OD (N=115) | Salmeterol 50 µg BID (N=116)
Nasopharyngitis (Infections and infestations) | 12 | 9 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 2 | 2
Headache (Nervous system disorders) | 5 | 10 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 2
Pyrexia (General disorders) | 0 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.